CLINICAL TRIAL: NCT03323229
Title: SatCare: Remote Support for Ambulance Clinicians in Medical Emergencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Scottish Ambulance Service (Unknown); NHS Highland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2-060-17
Record Dates: First submitted 2017-10-09; First posted 2017-10-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Emergency Medical Services; Emergency Service, Hospital
Keywords: Ultrasonography; Ambulances; Satellite Communications; Telemedicine
MeSH Terms: conditions — Emergencies | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Usual care (control group) (No Intervention): Patient receives care as usual.
- Enhanced communications & ultrasound (Experimental): The paramedic will record a brief video summary of the patient's condition, then remotely supported point of care ultrasound scans will be performed, and both file types sent to the hospital for review and feedback from the consultant.
  Interventions: Diagnostic Test: Enhanced communications & ultrasound

INTERVENTIONS:
Diagnostic Test: Enhanced communications & ultrasound — Paramedics will perform standardised point-of-care ultrasound scan protocols (specific to the patient's symptom set) and record a short (<1 minute) video summarising the patient's condition and current management. These will be transmitted via satellite to consultants at the receiving hospital before the ambulance leaves the incident scene. The emergency department consultants will provide support and advice on continuing patient management via standard ambulance communications systems while it is en route to the hospital.
  Arms: Enhanced communications & ultrasound

SUMMARY:
SatCare is a randomised controlled trial involving rapid standardised ultrasound assessment of patients with shock, major trauma, abdominal pain, chest pain or breathlessness in emergency ambulances. The scans will take less than 5 minutes and be transmitted to a hospital-based expert for review, providing support and instructions for optimal prehospital care.

Five Highland Scottish Ambulance Service ambulances covering areas more than 30 minutes from Raigmore Hospital, Inverness, UK, will be equipped with an ultrasound machine (M-Turbo, FujiFilm Sonosite) and satellite transmission system plus webcam, and will be deployed in real emergency situations. When dispatched to a potentially eligible patient, the attending paramedic will contact Raigmore Hospital's emergency department to check the availability of an emergency medicine specialist and obtain study group allocation (ultrasound with enhanced telecommunications plus usual care versus usual care alone). Following verbal consent from the patient, trained paramedics will perform the condition-specific scan protocol in the ambulance at the incident site, and transmit the recordings and patient video via satellite to the emergency department for specialist analysis. The consultant will give advice on patient management via standard ambulance communications systems while it is en route to the hospital.

The remotely supported prehospital ultrasound implementation will be examined in terms of its delivery and functioning. An economic evaluation will compare its use with care as usual for eligible patients transported by ambulance, modelling the costs and benefits of this service expansion and determining optimum use. It is hoped that the results, anticipated to be available in 2019, will provide an evidence base for the use of prehospital ultrasound for emergency care.

DETAILED DESCRIPTION:
Research objectives:

* To assess the patient health impact of enhanced telecommunications and remotely-supported point-of-care ultrasound scanning (RS-POCUS) in prehospital situations
* To assess the impact of introducing this intervention on current care systems, via interviews with various stakeholders involved in the trial (e.g., patients, paramedics, emergency medicine consultants, hospital management, etc.) and health economic modelling

Research questions:

* What is the health gain, as assessed by the EQ-5D-5L (EuroQol five dimension questionnaire, 5-level version) score at three months, associated with the use of enhanced telecommunications and RS-POCUS?
* What is the estimated cost-per-QALY associated with the prehospital RS-POCUS?
* Where in the care system and in which situations does the intervention produce the greatest impact?
* How does the use of RS-POCUS affect time to definitive treatment in the studied patient groups?

Patient Randomisation:

Patients will be randomized to the intervention or control group prior to obtaining consent (Zelen randomisation), an approach considered optimal in trials where care is time-critical and patients may be highly stressed. This simplifies and shortens the in-ambulance consent process because the details of the random allocation and its associated uncertainty don't need to be explained until later.

Randomisation is performed using randomisation envelopes with codes printed on them, located in the ambulances. Codes will be reported and recorded on the emergency department contact log when a potential patient call-out occurs. If on arrival at the emergency scene the patient meets the inclusion criteria, the paramedic will obtain the patient's study group allocation by opening the envelope.

Consent:

It is crucial that delays to patient transfer are reduced to an absolute minimum in the ultrasound scanning group. The process of scanning is rapid and offers virtually no risk to the patient, but delays due to requesting consent are potentially more problematic and need to be minimised as much as possible. It is therefore proposed to have a two-stage consent process: a brief verbal consent to scanning and data transmission in the ambulance, and on arrival at the hospital, full written consent to health record analysis and to complete a follow-up questionnaire three months later.

If patients are assessed by the paramedic to lack the mental capacity and understanding to provide meaningful consent, an eligible proxy (relative, welfare attorney or guardian) accompanying the patient may provide consent on his or her behalf in line with the Adults with Incapacity Act, Scotland (2000). If a participant who is unable to consent shows any signs of unwillingness to take part or distress, they will be immediately withdrawn from the study.

Patient follow-up:

Patients will be asked to complete a standard EQ-5D-5L (health-related quality of life) questionnaire 3 months after recruitment to the trial, plus a short satisfaction/service use questionnaire. Ten patients from both the scanned and control groups will be approached at this time to ask if they would be willing to be interviewed about the use of ambulance-based ultrasound. If other specific interesting themes meriting further investigation arise from the interviews, these may be explored further with additional interviews in other participants. Patient involvement in the trial will end on completion of this 3-month follow-up.

Analyses:

The primary outcome is defined as the patient EQ-5D-5L (EuroQol five dimension questionnaire) score three months after the original ambulance episode. Analysis will be on an intention to treat basis with a per protocol analysis as a sensitivity. Pre-specified descriptive subgroup analyses will examine EQ-5D-5L results by age group, reason for scan and transport distance.

The economic analysis will include both a within-trial economic evaluation and a model-based economic evaluation. The within-trial analyses will take the form of a cost-utility analysis from the perspective of the National Health Service. The model-based analysis will also take the perspective of the NHS, but try to take into account wider societal costs such as unpaid carer time and costs, using standard national figures to estimate these contributions. A Markov model will be used to extrapolate from the short-term trial outcomes into the longer term.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  * significant trauma: any case where the mechanism of injury, anatomical defect or physiological upset triggers the paramedic to pre-alert a 'trauma call' to the receiving Emergency Department
  * chest pain: pain felt below the clavicles and above the costal margin, whether anterior or posterior
  * shortness of breath: any patient complaining of 'shortness of breath' or with paramedic examination positive for 'respiratory distress' whether by increased respiratory rate, effort or both
  * abdominal pain: any pain felt below the costal margin and above the bony pelvis
  * cardiovascular shock of unknown origin: either a systolic blood pressure below 100 mmHg or any symptoms or signs of syncope on elevation of the head, cool peripheries or extended capillary refill time
* Attended by a study ambulance
* Recruitment occurs within the hours supported by the Emergency Department: Monday to Friday, 09:00 to 17:00

Exclusion Criteria:

* Non-emergency ambulance transfers
* General practitioner requested emergency ambulances
* Patients under arrest or held in prison
* No potential value in performing ultrasound (e.g., none of the diagnoses listed above)
* Lack of consent for scan (if in intervention arm)
* Lack of capacity to consent to scan / no patient representative to provide consent
* Evidence of any condition leading to lack of capacity to give informed consent prior to the commencement of the study, as documented on the patient's electronic patient record
* Non-English speakers
* Outside the emergency department supported hours (Monday to Friday, 09:00 to 17:00)
* Paramedic decision to exclude patient, for reasons such as urgency of transport (i.e., where thorough on-scene evaluation would not normally be offered) or other lack of suitability

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L (EuroQol five dimension, five level) score three months after the initial ambulance episode | 3 months post recruitment
  The EQ-5D-5L questionnaire includes assessments of mobility, self-care, daily activities undertaken, pain, discomfort, anxiety and depression.Completion of the EQ-5D-5L leads to the establishment of 243 distinct states, each with corresponding numerical quality of life value.

SECONDARY OUTCOMES:
Cost per QALY (Quality Adjusted Life Year) | 3 months post recruitment
  Estimates of cost per QALY are generated using costs and EQ-5D-5L score. The QALY is a measure of disease burden, encompassing both the quality and quantity of life lived. Quality of life is rated between 0 ('worst possible health') and 1 ('best possible health'). The QALY is calculated from the amount of time spent in a particular health state weighted by the utility (quality) score given to that health state.
  The QALY gained by a specific treatment is compared with an existing standard or no intervention. The relative costs of the two interventions are then compared and the cost of the new treatment in excess of the standard is calculated. This figure is then divided by the QALY of the new intervention to give the cost per QALY (£ per QALY). Lower costs per QALY are preferred by healthcare systems, as they are thought to provide better value for money.
Time from ambulance arrival at scene to definitive treatment or discharge | up to 3 months post recruitment
  Measured in hours and minutes
Mortality rate | up to 3 months post recruitment
Process evaluation (to investigate intervention use, acceptance and optimisation) | 15 months
  Includes interviews with stakeholders and anonymised descriptions of cases in which management was altered as a result of the intervention
Costs to the NHS | 15 months
  Covering staff and equipment costs, treatment costs, etc. Costs will be measured in UK Pounds Sterling and compiled into a Total Costs figure to compare costs with/without the intervention.
Relative efficiency calculations (cost-consequences analysis) | 15 months
  A cost-consequences analysis is an economic evaluation where disaggregated costs and a range of outcomes are presented to allow readers to form their own opinion on relevance and relative importance. A descriptive table presents the primary and secondary outcome results together with the estimates of the mean costs associated with each intervention.
Patient and staff satisfaction with the intervention | 15 months
  Collected using custom created questionnaires
Patient and staff satisfaction with the intervention | 15 months
  Collected using custom created interview schedules
Communications system connection speed | 15 months
  The communications system connection speed - the time to locate the satellite, connect to it, and connect to the end server - will be recorded (minutes and seconds). Any failure to connect will be noted.
Communications system data upload rate | 15 months
  Data upload speeds will be recorded (kb/s).

CONTACTS AND LOCATIONS:
Overall Officials: Leila Eadie, Principal Investigator — University of Aberdeen; Philip Wilson, Principal Investigator — University of Aberdeen
Locations (3):
- United Kingdom (3):
  - Centre for Rural Health, Inverness, Scotland
  - NHS Highland: Raigmore Hospital, Inverness, Scotland
  - Scottish Ambulance Service, Inverness, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eadie L, Mulhern J, Regan L, Mort A, Shannon H, Macaden A, Wilson P. Remotely supported prehospital ultrasound: A feasibility study of real-time image transmission and expert guidance to aid diagnosis in remote and rural communities. J Telemed Telecare. 2018 Oct;24(9):616-622. doi: 10.1177/1357633X17731444. Epub 2017 Sep 18. PMID 28920524
- See also: European Space Agency project website — https://business.esa.int/projects/satcare
- See also: University of Aberdeen project website — https://www.abdn.ac.uk/iahs/research/crh/projects/satcare.php